CLINICAL TRIAL: NCT02460302
Title: Vaginal Progesterone Versus Placebo for the Treatment of Vaginal Atrophy - a Double Blind Randomized Control Trial
Brief Title: Vaginal Progesterone Versus Placebo for the Treatment of Vaginal Atrophy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Inadequate staffing and funds
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Principal Investigator, Wendy Wolfman, Professor, Obstetrics and Gynaecology, University of Toronto, Mount Sinai Hospital, Canada
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12-0306-A
Record Dates: First submitted 2015-05-29; First posted 2015-06-02 (Estimated); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Atrophic Vaginitis; Menopause; Vulvovaginal Atrophy
MeSH Terms: conditions — Atrophic Vaginitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vaginal Progesterone (Experimental): In the experimental arm, the participants will be randomized (1:1 allocation) to receive a vaginal progesterone suppository (100mg) as the intervention.
  Participants will be instructed to insert the vaginal suppository into the vagina, as high as is comfortable for the patient. They are to insert the drug three days per week, on Monday, Wednesday and Fridays, preferably at bedtime. Patients will record the use of their medications. This will be done for the study period of 12 weeks.
  Interventions: Drug: Vaginal progesterone
- Placebo Comparator (Placebo Comparator): In the placebo arm, the participants will be randomized (1:1 allocation) to receive a vaginal suppository (100mg) containing hard fat without any active hormonal ingredient as the intervention.
  Participants will be instructed to insert the vaginal suppository into the vagina, as high as is comfortable for the patient. They are to insert the placebo three days per week, on Monday, Wednesday and Fridays, preferably at bedtime. Patients will record the use of their medications. This will be done for the study period of 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vaginal progesterone — Micronized vaginal progesterone 100mg inserted vaginally
  Other Names: Oripro
  Arms: Vaginal Progesterone
Drug: Placebo — Placebo suppository inserted vaginally
  Arms: Placebo Comparator

SUMMARY:
Atrophic vaginitis affects the majority of post-menopausal women. It is characterized by dryness and inflammation of the vagina, with thinning of the vaginal tissues. Atrophic vaginitis is caused by the decreased effect of estrogens post menopause. Traditionally, local estrogens have been used to treat atrophic vaginitis

Studies have shown that there are progesterone receptors in vaginal tissues. The use of progesterone to treat atrophic vaginitis has not yet been studied. However, its use has been studied in other populations including as a fertility medication in pregnant women.

There is a significant group of women who cannot use, choose not to use, or do not respond to estrogenic therapies. The goal of this study is to evaluate the efficacy of vaginal progesterone in the treatment of urogenital atrophy, compared to placebo. This study is a randomized, double-blind, placebo controlled trial. The ultimate goal is to expand the treatment options for patients with symptoms of vaginal atrophy.

DETAILED DESCRIPTION:
Introduction

Atrophic vaginitis is a condition that affects the majority of postmenopausal women. It is characterized by dryness and inflammation of the vagina, with thinning of the vaginal tissues. Atrophic vaginitis is caused by the decreased effect of estrogens post menopause. This condition becomes more significant over time, as systemic levels of estrogen decline. This is in contrast to vasomotor symptoms of the peri-menopause and early post-menopause, which generally subside as time passes. Therefore, because of an aging demographic, it is a condition that will have an ever-growing population requiring its treatment. However, only a minority of women that suffer from atrophic vaginitis seek medical help. Instead, many women make difficult lifestyle changes to deal with their symptoms. This may include avoiding sexual activity to avoid the associated pain with intercourse.

The vagina has a significant of estrogen receptors. Effects of estrogens on the vagina have been well studied. Currently, there are numerous estrogenic therapy options, both systemic and local, to treat symptoms of vaginal atrophy. Recent evidence supports the efficacy of this population of lower vaginal estrogen doses (10mcg) than previously used (25mcg). Emerging evidence is demonstrating efficacy for ultra-low doses of estrogen therapies. The search for such low doses of estrogen therapy suggests an ongoing distrust among both the public and the scientific community for the acceptability of estrogen therapy. Despite these lower does, many women are still unable or unwilling to use local estrogen therapy. The options for such women are limited.

Studies have shown that there are progesterone receptors in vaginal tissues. The use of progesterone to treat atrophic vaginitis has not yet been studied. However, its use has been studied in other populations. Progesterone therapy has long been used to support fertility in reproductive aged women, with few side effects. Progesterone also has a long history of use in the menopausal population. It is administered as combined therapy with estrogen, providing endometrial protection against hyperplasia and malignancy. This addition of a progestin to systemic estrogen therapy for women with a uterus is the standard of care.

There is a significant group of women who cannot use, choose not to use, or do not respond to estrogenic therapies. The goal of this study is to evaluate the efficacy of vaginal progesterone in the treatment of urogenital atrophy, compared to placebo. The ultimate goal is to expand the treatment options for patients with symptoms of vaginal atrophy.

Hypothesis

The current standard of care for women with vaginal atrophy is treatment with local estrogen. However, a significant number of women cannot or prefer not to use estrogen therapy because of potential side effects. The alternative options are few and provide limited symptomatic relief. The investigators propose vaginal progesterone as an alternative therapeutic option for the relief of vaginal atrophy.

The objective of the study is to find and effective alternative therapeutic option to vaginal estrogen, in the way of vaginal progesterone, for the treatment of vaginal atrophy.

Hypotheses include:

1. Local progesterone will be superior to placebo for patient reported symptoms.
2. Women receiving a course of local progesterone will have superior physician assessment of vaginal atrophy compared to placebo.
3. Local progesterone will improve vaginal pH and maturation index compared to placebo.

Methods

Population:

The study will be conducted out of Dr. Wolfman's Gynecology and Menopause Clinics at the Mount Sinai Hospital Ontario Power Generation Building. Women who are post menopausal and presenting with complaints of vaginal atrophy will be eligible for inclusion in the study. Women may self identify to participate in the study, in response to recruitment materials present in the clinical office, or may be identified by their health care professional.

Study Design

This will be a randomized, double blinded, placebo controlled trial. The participants will be randomized on a 1:1 ratio to either vaginal progesterone suppository, or an identical placebo. The dose of the vaginal progesterone suppository is 100mg.

The study medication will be provided by the Australia Research Centre for Health of Women and Babies, University of Adelaide.

Randomization will be completed by a computer generated system through the Mount Sinai Pharmacy. Study medications will be shipped directly to the homes of study participants.

Participation in the study will consist of two clinical visits. The first clinical visit is a baseline visit. The second visit will occur following twelve weeks of using the study medication. The visits will be similar in procedures and time involved, as follows:

Baseline:

* Symptom questionnaire
* Clinical breast exam
* Vaginal speculum exam, including a Pap test
* Serum progesterone level
* Cholesterol panel, if not completed within previous year
* Approximately 60 minutes in length

Follow-Up:

* Symptom questionnaire
* Clinical breast exam
* Vaginal speculum exam, including a vaginal exam
* Serum progesterone level
* Approximately 60 minutes in length

The symptom questionnaire will ask patients to rate their symptoms of vaginal atrophy. It will evaluate the following:

* vaginal dryness
* vaginal and/or vulvar irritation or itching
* vaginal pain associated with sexual activity Symptoms will be rated on a scale of 0 through 3, with zero being none, one being mild, two being moderate and three being severe. Patients will be asked to identify their most bothersome symptom. Patients who are not sexually active may participate.

The vaginal exam will be performed by the study gynecologist, Dr. Wolfman or the Menopause fellow.

Patients will also have a vaginal speculum exam performed by the staff gynecologist or fellow. Vaginal swabs will be collected to assess vagina pH and maturation index. pH will be measured by inserting a pH test strip into the upper third of the vagina and completing the reading while the strip is damp. A sample slide with vaginal cells will be collected to be sent to the laboratory in order to measure maturation value.

Clinical breast exam will be conducted to rule out any clinically evident breast disease prior to the study, and following the 12 weeks of study participation.

Blood work will be collected to assess serum progesterone levels. The investigators anticipate systemic absorption to be low. A serum cholesterol panel will also be collected to ensure the patient has normal baseline values if there is not a recent (within one year) result available.

Adverse events will also be recorded outcomes. These include headaches, vaginal discharge, vulvo-vaginal mycotic infection (either diagnosed or self-treated), increased vulvo-vaginal pruritis, vaginal bleeding and other. On the Consent Form, there is contact information for patients so they are able to reach study personnel, should they have any questions or concerns, or need to report adverse events. A 24 hour emergency number is also available to patients in the study, should they need to contact study personnel at any time. Adverse events will be dealt with on a case-by-case basis, as they occur. A record will be made of any and all adverse events, by the study investigators. For any serious adverse events, the patients will be advised to immediately study the study medication. Unblinding of the staff and/or study participants will occur when this is deemed necessary.

All relevant clinical outcomes will be evaluated before therapy initiation, at the baseline visit, and following 12 weeks of therapy. Improvement in symptoms between the two time periods will be evaluated.

ELIGIBILITY:
Inclusion criteria:

1. Age greater than or equal to 45, unless the patient has had a bilateral oophorectomy
2. Amenorrheic for greater than one year and/or FSH > 40IU/mL
3. Women who have had a bilateral oophorectomy will be eligible at any age
4. Patients must have greater than or equal to two urogenital atrophy symptoms:

   * vaginal dryness
   * vaginal irritation
   * vaginal soreness
   * dyspareunia

Exclusion criteria:

1. Age less than 45
2. Systemic or local hormone replacement therapy use within three months of entry into study
3. Known or suspected history of breast cancer
4. Hormone dependent tumor
5. Genital bleeding of unknown cause
6. Current vaginal infection requiring treatment
7. Known allergy to test constituents
8. Serious disease or chronic condition that could interfere with compliance
9. Active thrombophlebitis, or history of a hormone-associated thrombophlebitis
10. Kidney disease
11. Liver dysfunction or disease
12. High LDL levels

Women who have used systemic or local hormone replacement therapy will be ineligible for participation in the study. If these women wish to participate, they must undergo a washout period. This would be as follows:

* eight weeks for oral estrogen and/or progestin therapy
* four weeks for transdermal or local vaginal hormone therapies
* eight weeks for progestin containing intrauterine system

Participants who are completing a washout period must complete the study questionnaire following the washout period.

Women will not be allowed to continue or commence use of non-hormonal therapies, including vaginal moisturizers, while they are in the study, However, we will allow the use of vaginal lubricants for sexual intercourse. Their use will be recorded on the patient questionnaire.

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-12 (Estimated); Primary Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Perceived Improvement in most bothersome vulvovaginal symptom | 12 weeks
  Improvement in patient-identified most bothersome symptom (vaginal dryness, itching, soreness, pain with sexual activity)

SECONDARY OUTCOMES:
Change in physician-assigned vaginal health index score based on a detailed rating scale | 12 weeks

OTHER OUTCOMES:
Change in vaginal maturation index value | 12 weeks
Change in vaginal pH values | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Wendy L Wolfman, MD, FRCSC, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Lara LA, Cartagena-Ramos D, Figueiredo JB, Rosa-E-Silva ACJ, Ferriani RA, Martins WP, Fuentealba-Torres M. Hormone therapy for sexual function in perimenopausal and postmenopausal women. Cochrane Database Syst Rev. 2023 Aug 24;8(8):CD009672. doi: 10.1002/14651858.CD009672.pub3. PMID 37619252